CLINICAL TRIAL: NCT02591745
Title: International Fetal Anesthesia Database
Acronym: iFAD
Status: Active, not recruiting | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other); Universitaire Ziekenhuizen KU Leuven (Other); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Titilopemi Aina, MD MPH, Associate Professor, Baylor College of Medicine
Other Study IDs: H- 35126
Record Dates: First submitted 2015-10-28; First posted 2015-10-30 (Estimated); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Determination of Neurological Outcomes
Keywords: Fetal; Anesthesia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Fetal intervention — Type of fetal conditions requiring intervention and medications administered to fetuses undergoing varying types of fetal intervention will be documeted in this database.

SUMMARY:
This registry aims to gather anesthetic medications administered to fetuses directly as well as those administered via the mother during fetal intervention procedures. The goal is to assesss short and medium term outcomes as well as long term outcomes of these babies whao have received medication in utero. The long term outcomes will include but are not limited to neurodevelopmental outcomes.

DETAILED DESCRIPTION:
Advances in technology have allowed for an increase in procedures performed on the fetus in utero; these procedures involve the administration of different anesthetics (sedative- hypnotic agents and or volatile agents) to the mother and sometimes directly to the fetus in order for succesful completion of the procedure. Very few instiututions in the world perform these procedures in any significant number. The establishment of this database will serve to consolidate information regarding anesthetic drugs administered for these procedures, thereby helping to establish best practice guidelines, determine medium and short term outcomes or complications and also facilitate long term neurodevelopmental assessment of children that have undergone these procedures in utero with 5 and 10 year neurodevelopmental assessment.

ELIGIBILITY:
Inclusion Criteria: Pregnant women, fetuses and children

Exclusion Criteria: Non-pregnant women

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Mothers whose fetuses require fetal intervention for a variety of conditions. Fetuses who have undergone surgical intervention while in-utero.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Fetal complications | Peri-operative
  resuscitation efforts during surgery or peri-operative demise

SECONDARY OUTCOMES:
Maternal hypotension or other maternal complications | Peri-operative period

CONTACTS AND LOCATIONS:
Overall Officials: Titilopemi Aina, M.D., M.P.H., Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Baylor College of Medicine, Houston, Texas, United States